CLINICAL TRIAL: NCT00535756
Title: One Week Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multi-Center Study With Creon® 25000 Minimicrospheres™ in Subjects With Pancreatic Exocrine Insufficiency After Pancreatic Surgery, Followed by an Open-Label Long-Term Extension of 1 Year
Brief Title: Creon After Pancreatic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Products (Industry)
Collaborators: Quintiles, Inc. (Industry); Data Map GmbH (Unknown)
Responsible Party: Gregor Eibes/Clinical Trial Manager, Abbott Products
Organization: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S245.4.008; 2005-004854-29 (EudraCT Number)
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Pancreatic Insufficiency
Keywords: Pancreatic Exocrine Insufficiency After Pancreatic Surgery
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Creon
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Creon — 3 capsules Creon with 25000 lipase units per main meal (3 main meals) plus 2 capsules per snack (2-3 snacks)
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
This study will provide efficacy data for Creon 25000 MMS in PS patients as well as long-term safety data. During the long-term treatment with Creon 25000 nutritional parameters will be assessed and correlated with CFA

ELIGIBILITY:
Inclusion Criteria

Pancreatic exocrine insufficiency has to be proven (in medical history) by the following criteria:

* Direct or indirect pancreatic function test (except stool fat excretion) and
* Steatorrhoea: stool fat > 15 g/day (using van de Kamer method)
* Proven chronic pancreatitis
* Females of child-bearing potential must agree to continue using a medically acceptable method of birth control

Exclusion Criteria

* Subjects in an unstable situation (catabolic) after pancreatic surgery
* Ileus or acute abdomen
* Current excessive intake of alcohol or drug abuse
* Hypersensitivity vs porcine proteins / pancreatin
* Subjects taking digestive enzyme preparations have to stop them before start of the run-in period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in CFA from baseline to the end of double blind treatment | 7 days after baseline

SECONDARY OUTCOMES:
CNA, stool fat, stool weight, nutritional parameters, clinical symptomatology, SF-36, BMI | 7 days after baseline, and end of open-label period (1 year of open label treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Guenter Krause, MD, Study Director — Abbott Products
Locations (15):
- Bulgaria (2):
  - Site Reference ID/Investigator# 45022, Rousse
  - Site Reference ID/Investigator# 45020, Sofia
- Germany (4):
  - Site Reference ID/Investigator# 45026, Greifswald
  - Site Reference ID/Investigator# 45025, Hamburg
  - Site Reference ID/Investigator# 45027, Heidelberg
  - Site Reference ID/Investigator# 45024, Munich
- Hungary (6):
  - Site Reference ID/Investigator# 45126, Békéscsaba
  - Site Reference ID/Investigator# 45121, Budaörs
  - Site Reference ID/Investigator# 45127, Dunaújváros
  - Site Reference ID/Investigator# 45115, Gyula
  - Site Reference ID/Investigator# 45116, Sopron
  - Site Reference ID/Investigator# 45114, Szeged
- Italy (3):
  - Site Reference ID/Investigator# 45130, Bologna
  - Site Reference ID/Investigator# 45129, Padua
  - Site Reference ID/Investigator# 45128, Verona